CLINICAL TRIAL: NCT00667030
Title: Aging, Lifestyle and Inflammation in Veterans Exercising
Acronym: ALIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jacob Blumenthal, GRECC Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00041199
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Inflammation; Aging; Metabolism; Exercise
Keywords: Inflammation; Aging; Metabolism; Exercise
MeSH Terms: conditions — Inflammation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Modification (Experimental): Combined hypocaloric diet and aerobic exercise training
  Interventions: Behavioral: Weight loss and aerobic exercise training

INTERVENTIONS:
Behavioral: Weight loss and aerobic exercise training — Weight loss and aerobic exercise training

SUMMARY:
Over half of adults in this country are overweight. This increases risk for heart and blood pressure problems, cancer, stroke and arthritis. While it is difficult to lose large amounts of weight and keep it off, even small amounts of weight loss can improve health. Furthermore, fat is increasingly recognized as a source of substances that increase inflammation. It may be that some of the adverse consequences of being overweight are due to increased inflammation. We are asking you to volunteer for a research study in which you may lose a moderate amount of weight and increase your activity. It is important that you read and understand the information on this form.

The purposes of these studies are to determine the influence(s) of age and body composition on the production of inflammatory chemicals by fat (adipose tissue), the mechanisms controlling this, and if a weight loss and aerobic exercise intervention results in a decrease in inflammation.

DETAILED DESCRIPTION:
Adipose tissue is increasingly recognized as more than an inert depot serving not only to accept and store excess energy in the form of triglycerides, but also to secrete hormones and adipokines that have substantial effects on lipid and glucose metabolism. Furthermore, there are depot differences in metabolic function, as well as adipokine content. However, the physiology both underlying and consequential to these observations remains unknown. This research is therefore designed to examine:

1) the effects of aging and obesity on regional adipokine secretion and expression, 2) whether elevated adipokine levels in older obese people are due to increased macrophage infiltration into subcutaneous adipose tissue and/or related to total, subcutaneous or visceral abdominal fat (SAT or VAT) distribution, and 3) the relationship of adipokines to insulin resistance and the constituents of the metabolic syndrome.

Specifically, we aim to determine:

1. if the expression and secretion of a) the inflammatory markers SAA, IL-6, TNF-a, MCP-1 is greater, and b) the anti-inflammatory hormone adiponectin is lower in SC abdominal and gluteal adipose tissue from older, compared to middle-aged and younger obese subjects across a narrow range of obesity and waist circumference;
2. if these age-associated changes in adipokine production are a)due to the degree of macrophage infiltration of regional adipose tissue, and/or differences in a greater degree of visceral and/or differences in ABD fat distribution (SAT, VAT), and b) related to glucose and lipid metabolic profiles of the subjects; and
3. the effects of a WL+AEX intervention on regional adipokine expression and secretion, circulating levels of CRP and the above adipokines, and glucose and lipid metabolism in a subset of obese sedentary individuals with greater than two components of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-40 kg/m2
* Waist 80-120cm (men), 70-110cm (women)
* Stable Medical Regimen > or = 30 days
* All women over the age of 50 must be postmenopausal for at least 1 year, have serum FSH >30 mIU/ml, and agree to remain off hormone replacement therapy for the duration of the study

Exclusion Criteria:

* Pregnancy or Nursing Mothers
* Cigarette Smoking
* Diabetes on Medication or Fasting Glucose >126 mg/dl
* Poorly controlled hypertension requiring >3 drugs or beta blockers
* Hyperlipidemia with TG>400mg/dl, LDL>190mg/dl or on Lipitor or Crestor
* Other medications affecting glucose, lipid or cytokine levels
* Thyroid Disease
* Weight gain/loss >5kg in preceding 3 months
* Alcohol >3oz/day
* Caffeine >120 oz/day
* Chronic liver, renal or hematological disease
* Lung disease requiring oxygen
* Active cancer on radiation or chemotherapy treatment
* HIV (+) or other disease prone to malnutrition
* Sickle cell anemia
* Active psychosis or dementia
* Chronic untreated depression
* Hemiparetic Stroke
* Coronary Artery or cerebrovascular disease precluding exercise
* Implantable defibrillator
* Other medical condition precluding exercise testing or participation in exercise and weight loss programs, as per medical judgement of study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Regional Adipokine Release | 6 month

SECONDARY OUTCOMES:
Cardiovascular Fitness Body Composition Glucose Tolerance/Insulin Sensitivity | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jacob B Blumenthal, MD, Principal Investigator — Baltimore VA Medical Center, University of Maryland
Locations (1):
- University of Maryland; Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No